CLINICAL TRIAL: NCT06380010
Title: Optimizing Dietary Habits in Adolescents With Polycystic Ovary Syndrome: Personalized Mediterranean Diet Intervention Via Clinical Decision Support System. A Randomized Controlled Trial
Brief Title: Mediterranean Diet Intervention in Adolescents With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iaso Maternity Hospital, Athens, Greece (Other)
Collaborators: Harokopio University (Other); University of Peloponnese (Other)
Responsible Party: Principal Investigator, Panos Papandreou, Maria Skouroliakou, Associate of Professor in Harokopio University of Athens, Iaso Maternity Hospital, Athens, Greece
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IASO HOSPITAL (ATHENS-GREECE)
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: Recruitment involved adolescents with polycystic ovary syndrome. Participants, who expressed their willingness to take part, attended personal meetings with the appointed dieticians who provided comprehensive explanations on the objectives, methods, and the potential benefits/risks of the study. A leaflet with related information was provided to all patients. Every eligible volunteer, and their guardian, signed a written informed consent and then kept a hard copy of the signed document. All eligible females were recruited in 12/2019 and were randomly allocated in groups of one to either the Control group (CG) or the Intervention group (IG). The IG received a personalized Mediterranean dietary plan, delivered through a clinical decision support system, while the CG received general dietary advice. Every participant had two individual sessions with the assigned dietician, at the beginning and at the trial endpoint, which involved anthropometry, dietary assessment, and blood withdrawal.
Who Masked: Outcomes Assessor
Masking Description: Treatment allocation was not revealed to the appointed statistician until the end of the study and release of the final outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Each participant was assigned to a highly skilled dietician. The dietician implemented an individualized daily dietary regimen according to the Mediterranean diet produced by the clinical decision support system (CDSS) software. The CDSS was utilized to calculate all necessary components for the synthesis of the dietary plan, which was renewed every 15 days. Participants of the Intervention group obtained unique login credentials for the CDSS and received instruction on its operation from the designated dietitians. They were directed to access their CDSS account remotely on a weekly basis in order to monitor their nutritional status (body weight and healthy eating) and to complete a three-day dietary journal; this information was automatically accessible to the dietitians. Telephone interviews were conducted every other week in order to supplement the nutritional and lifestyle consultations. In addition, unanticipated phone calls requesting 24-hour dietary recalls were received.
  Interventions: Other: Mediterranean diet group
- Control Group (No Intervention): The Control group participants were not provided with CDSS. They simply got basic lifestyle instructions based on the "National Dietary Guidelines for Children and Adolescents" during phone call sessions with the dieticians every 15 days. The ladies in the Control group were directed to maintain a food diary for three consecutive days each week, which they then transmitted to the designated dietician via email. Once again, unsolicited phone calls were conducted in order to acquire 24-hour dietary recalls.

INTERVENTIONS:
Other: Mediterranean diet group — Females who met the inclusion and exclusion criteria were allocated in groups of one to either the Control group or the Intervention (MD) group using a random assignment method applied by an independent statistician. During the trial, every participant in both groups had two individual sessions with the assigned researchers. These sessions took place at the beginning of the trial and three months later, and involved anthropometry measurements, evaluation of dietary habits, assessment of psychological well-being, and collection of blood samples. Treatment allocation was not revealed to the appointed statistician until the end of the study and release of the final outcomes.
  Arms: Intervention Group

SUMMARY:
The aim of the present randomized controlled study was to examine wether a clinical decision support stystem would increase the adherence to the Mediterranean diet (MD) of adolescent girls, aged 15-17 years, diagnosed with polycystic ovary syndrome. The intervention lasted for 3 months and in total, 40 girls were randomly assigned to either the MD group (n=20) or a Control group receiving general nutritional advice (n=20). Anthropometry, nutritional intake, psychological well-being, and blood markers were analyzed at the begninning and the end of the trial.

DETAILED DESCRIPTION:
The aim of the present randomised controlled trial was to investigate the effects of a Mediterranean Diet (MD) intervention delivered through a Clinical Decision Support System (CDSS) on various dietary, health parameters and anxiety in adolescent females, aged 15-17 years, with PCOS. A randomized controlled trial was conducted with 40 adolescent females diagnosed with PCOS, randomly assigned to either an Intervention group (IG) (n=20) or a Control group (CG) (n=20). The IG received personalized dietary guidance based on the MD principles, delivered through a CDSS, while the CG received general nutritional advice. Measurements of dietary intake, anthropometric indices, biochemical markers, and psychological well-being were collected at baseline and after a 3-month intervention period. After 3 months, significant improvements were observed in the IG compared to the CG. Adherence to the MD increased significantly in the IG, leading to decreased caloric intake, fat, saturated fatty acids, and dietary cholesterol, and increased intake of monounsaturated fatty acids. Conversely, the CG experienced an increase in fat and dietary cholesterol intake. Both groups exhibited an increase in fiber intake, with a more pronounced rise observed in the MD group. Psychological well-being showed a significant reduction in anxiety levels in the IG group, while no significant change was observed in the CG. The intervention led to improvements in dietary patterns, body composition, and psychological well-being. These results underscore the importance of dietary interventions tailored to the MD principles in the management of PCOS among adolescent females.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed with PCOS females <18 years of age.
2. Females with guardians who provided signed participation consent.

Exclusion Criteria:

1. Females ≥18 years of age.
2. Females suffering from severe illnesses (i.e., organ failure, autoimmune diseases, congenital metabolic disorders), psychiatric disease or with emerging health issues that could hinder the trial.
3. Pregnant or lactating females.
4. Females diagnosed with alcoholism or drug addiction.
5. Females being under any drug treatment.
6. Females followed a specific type of diet within the past 5 years or have used nutrient or non-nutrient supplements within the last 6 months.
7. Females with guardians non able to read and understand the consent information.

Ages: 15 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — sex was biologically identified
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Adherance to the Mediterranean diet | 3 months
  Adherance was assessed with the Kidmed score

SECONDARY OUTCOMES:
Improvement of psychological well-being | 3 months
  Psychological well-being was assessed by the Hospital Anxiety-Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Locations (1):
- IASO Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foscolou A, Papandreou P, Gioxari A, Skouroliakou M. Optimizing Dietary Habits in Adolescents with Polycystic Ovary Syndrome: Personalized Mediterranean Diet Intervention via Clinical Decision Support System-A Randomized Controlled Trial. Children (Basel). 2024 May 24;11(6):635. doi: 10.3390/children11060635. PMID 38929215